CLINICAL TRIAL: NCT02401295
Title: An Open-Label Phase I Trial to Evaluate the Safety and Tolerability of ATRA, Celecoxib, and Itraconazole Administered As Maintenance Treatment Post-Autologous Transplantation in Relapsed Multiple Myeloma
Brief Title: ATRA, Celecoxib, and Itraconazole as Maintenance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Guido Tricot, Principal Investigator, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201311791
Record Dates: First submitted 2015-03-18; First posted 2015-03-27 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Relapsed Multiple Myeloma
Keywords: Relapsed multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Tretinoin; Celecoxib; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ATRA/celecoxib/itraconazole (Experimental): All maintenance drugs will be given on days 1-21 of each cycle, followed by 14 days off treatment. Cycles will be repeated every 35 days (+/- 3 days) for a total of five cycles.
  Each patient enrolled will receive ATRA 20mg twice per day by mouth. Dose modifications are not allowed unless excessive toxicity occurs. In this case, ATRA will be de-escalated by 50% to 10mg twice per day by mouth.
  The dose of celecoxib for all patients enrolled will be 400 mg twice per day by mouth. If creatinine level increases to more than 2 mg/dl and cannot be corrected by increased oral fluid intake or other measures, the dose of celecoxib will be decreased by 50%. If creatinine level does not drop below 2 mg/dl on the reduced dose, celecoxib will be discontinued.
  The dose of itraconazole for all patients enrolled will be 200 mg twice per day by mouth. Dose modifications are not allowed.
  Interventions: Drug: ATRA; Drug: Celecoxib; Drug: Itraconazole

INTERVENTIONS:
Drug: ATRA
  Other Names: All-Trans-Retinoic Acid; tretinoin
Drug: Celecoxib
  Other Names: Celebrex
Drug: Itraconazole
  Other Names: Sporanox; Onmel

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability associated with the combination of ATRA/celecoxib/itraconazole as maintenance therapy given after an autologous stem cell transplant in relapsed multiple myeloma patients.

DETAILED DESCRIPTION:
Primary objective:

To evaluate safety and tolerability associated with the combination of ATRA/ celecoxib/itraconazole given after a salvage transplant for relapsed myeloma in 25 patients in a cycle schedule consisting of three weeks of treatment followed by a rest period of two weeks for a total of five cycles. Subjects will be evaluable only if they have received at least one dose of maintenance treatment. The salvage transplant is not part of this study.

Secondary objective:

To explore changes in frequency and molecular signature in the multiple myeloma stem cell (MMSC) fraction based on flow-cytometric assays and gene expression profiling before and after the experimental treatment and to correlate outcome with expression levels of RARα2 at time of relapse.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsed multiple myeloma
* Recent salvage transplant (≤ 6 months but ≥ 45 days post-transplant prior to study enrollment) for relapse
* 18-75 years of age at the time of study entry
* Platelet count ≥70K/mm3 un-transfused
* Resolution of all transplant-related toxicity to ≤ grade 2 per CTCAE v.4
* Left ventricular ejection fraction as measured by ECHO or MUGA should be ≥ 40%
* Creatinine of ≤ 2 mg/dl and a calculated GFR of >50mL/min/1.73m2
* A total bilirubin, ALT, AST, and alkaline phosphatase of ≤ 2 ULN
* Performance status of 0-2 based on the ECOG criteria. Patients with performance status 3 or 4, based solely on bone pain, are also eligible, provided that there is a source document to verify this
* Prospective study participants must be informed of the investigational nature of the study and must have signed an IRB-approved informed consent form in accordance with institutional and federal guidelines

Exclusion Criteria:

* Prior allogeneic transplant
* Greater than grade 2 motor neuropathy or greater than grade 3 sensory neuropathy at screening
* Uncontrolled diabetes
* Recent (< 6 months) myocardial infarction, unstable angina, CABG or stent placement in the last 2 years, difficult-to-control congestive heart failure, uncontrolled hypertension (systolic blood pressure > 160 mm or a diastolic BP > 110 mm under normal conditions and while on appropriate anti-hypertensive medications), or difficult- to-control cardiac arrhythmias
* Evidence of QT prolongation and/or torsades de pointes (TdP) on EKG.
* Any co-morbid condition that poses a greater threat to the patient's life expectancy than the recurrent myeloma
* No concurrent malignancy with a life expectancy of less than two years, or one that requires ongoing chemotherapeutic intervention at screening
* Presence of an infection that requires intravenous antibiotics
* Pregnant or nursing females. Any patient of reproductive potential may not participate unless he/she has agreed to use an effective contraceptive method as covered during the informed consent process
* Known history of an HIV seropositive test

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety | 6 months

SECONDARY OUTCOMES:
Blood and Bone Marrow Aspirate Samples as a measure of changes to the MMSC (multiple myeloma stem cell) fraction. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Guido Tricot, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States